CLINICAL TRIAL: NCT01058512
Title: A Phase 2 Trial of NOV-205 in Chronic Viral Hepatitis C Patients (Genotype 1) Who Have Failed Treatment With Pegylated Interferon Plus Ribavirin
Brief Title: A Trial of NOV-205 in Hepatitis C Patients Who Failed Standard Therapy
Acronym: NOV-205
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cellectar Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOV205-C201
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis C
Keywords: hepatitis C; chronic HCV; viral HCV; genotype 1; failed treatment with pegylated interferon plus ribavirin
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single (Experimental): single-arm study
  Interventions: Drug: NOV-205

INTERVENTIONS:
Drug: NOV-205 — There will be 4 treatment Groups with 10 patients in each group:
  * Group A: 30 mg NOV-205 daily subcutaneous administration for 49 days
  * Group B: 30 mg NOV-205 daily subcutaneous administration for 98 days
  * Group C: 60 mg NOV-205 daily subcutaneous administration for 49 days
  * Group D: 60 mg NOV-205 daily subcutaneous administration for 98 days

SUMMARY:
The purpose of this research study is to find out the effect of the investigational drug NOV-205 on the level of hepatitis C virus in the blood and whether NOV-205 is well-tolerated at different doses when taken by subjects with hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* A serum HCV RNA level of >100,000 IU/ml using a quantitative, branched-chain-DNA (bDNA)-based assay (lower limit of quantitation = ~650 IU/ml) or other equally sensitive quantitative methods.
* Infection with genotype 1 HCV
* Documented failure to respond to treatment (defined as a patient who did not achieve an early viral response (EVR) (≥2 log reduction in serum HCV RNA or undetectable HCV RNA after 12 weeks of treatment) OR is serum HCV RNA positive after 24 weeks of treatment with pegylated interferon plus ribavirin for hepatitis C
* Adequate laboratory parameters
* Women of childbearing potential willing to use two acceptable methods of birth control during trial participation or are sterile or post-menopausal (defined as not having a menstrual cycle for greater than two years)
* Sexually active male subjects are practicing acceptable methods of contraception during trial participation
* Have the ability to understand the requirements of the trial, have provided written informed consent, and agree to abide by the trial restrictions and to return for the required assessments
* The subject must be able to self administer daily subcutaneous injections or their caregiver must be able to administer daily subcutaneous injections

Exclusion Criteria:

* Clinical, laboratory, or histological evidence of liver cirrhosis
* Evidence of hepatic decompensation (presence of or a history of ascites, hepatic encephalopathy, variceal bleeding, or hepatocellular carcinoma)
* Co-infection with human immunodeficiency virus (HIV) or active hepatitis B virus (HBV) (as determined by presence of hepatitis B surface antigen (HBsAg)
* Have received pegylated interferon and/or ribavirin within the 60 days prior to enrollment
* Any known preexisting medical condition that could interfere with the subject's participation in and completion of the protocol
* Pregnant female or nursing mother

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To evaluate changes in viral load | 16 months
To evaluate changes in serum ALT and AST levels | 16 months
To evaluate the durability of any changes in viral load and serum ALT and AST | 16 months
To establish the safety profile of NOV-205 | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Koff, MD, Principal Investigator
Locations (6):
- United States (6):
  - Borland-Grooover Clinic, Jacksonville, Florida
  - Venture Research Institute, LLC, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - MetroWest Medical Center, Framingham, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina